CLINICAL TRIAL: NCT05013645
Title: Evaluation of Skin Hydration in Adults With Dry Skin Using a Moisturizer With an Added Sterilized Probiotic
Acronym: DAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Dermatology Associates of Tallahassee (Unknown); Quorum Innovations (Unknown)
Responsible Party: Principal Investigator, Sharon Liebrich, Institutional Representative, Florida State University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FSUIRB0188
Record Dates: First submitted 2021-08-05; First posted 2021-08-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dry Skin
Keywords: Probiotic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterilized probiotic (LfQi601) (Experimental): Sterilized probiotic topically administered.
  Interventions: Other: Sterilized probiotic LfQi601
- Gel control product (Placebo Comparator): Inactive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Sterilized probiotic LfQi601 — Sterilized probiotic topically administered.
  Arms: Sterilized probiotic (LfQi601)
Other: Placebo — Gel control product
  Arms: Gel control product

SUMMARY:
Double-blind placebo-controlled clinical trial to evaluate the effectiveness of a sterilized probiotic on skin health and hydration in adults with dry skin.

The goal of the study is to determine if the addition of a skin-conditioning probiotic to a standard gel product will moisturize the skin, support a healthy skin microbiome, and be readily tolerated by adults with dry skin.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability to attend study visits for the duration of the study
3. English-speaking
4. 18-90 years of age
5. Score of a 2 or higher in one of the four areas assessed on the Dry Skin Area and Severity Index (DASI)

Exclusion Criteria:

1. Current self-reported pregnancy or active intent to conceive
2. Current lactation
3. Fever within 7 days of study enrollment
4. Self-reported use of systemic antibiotics (oral or injectable) in the past 6 weeks.
5. Any clinically significant medical or psychological disorder, condition, or disease that in the opinion of the investigator exposes the subject to unacceptable risk by participating in the study or interferes with the subject's ability to complete the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Corneometer Measurements | Study Days 1, 14, 28, 35
  Measures change in skin surface hydration at study days 1, 14, 28 and 35
Tewameter Measurements | Study Days 1, 14, 28, 35
  Measures change in rate of skin surface water loss at study days 1, 14, 28, 35

SECONDARY OUTCOMES:
Skin microbiome analysis | Study Days 1, 28
  Changes in the composition (abundance and diversity) of skin lesional microbiome communities between Days 1 and 28 as demonstrated by genomic region amplification and analysis of sterile skin swab sample using standard protocols to compare associated organisms between the 2 time points
Change in Skindex16 Quality of Life over study days 1, 14, 28, 35 | Study Days 1, 14, 28, 35
  Symptom-based scoring tool
Change in Dry Skin Area and Severity Index (DASI) between study days 1 and 28 | Study Days 1, 28
  Symptom-based scoring tool
Change in Dryness Self Assessment (D-VAS) over study days 1, 14, 28 and 35 | Study Days 1, 14, 28, 35
  Symptom-based scoring tool
Change in Itchiness Self Assessment (I-VAS) over study days 1, 14, 28 and 35 | Study Days 1, 14, 28, 35
  Symptoms-based scoring tool

CONTACTS AND LOCATIONS:
Overall Officials: Eva Berkes, MD, Principal Investigator — Florida State University College of Medicine and Quorum Innovations
Locations (1):
- Dermatology Associates of Tallahassee, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No